CLINICAL TRIAL: NCT00391469
Title: Study of the Use of Mild Hypothermia in Out-of-hospital Cardiac Arrest Using a Rapid Infusion of 2 Liters of Cold Normal Saline
Brief Title: Induction of Mild Hypothermia Following Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Medic One Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Francis Kim, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29121-B; R01HL089554 (NIH)
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: cardiac arrest; mild hypothermia
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- control treatment (No Intervention)
  Interventions: Other: Rapid infusion of 2 liters of 4oC normal saline; Drug: Rapid infusion of cold normal saline

INTERVENTIONS:
Other: Rapid infusion of 2 liters of 4oC normal saline — Patients randomized to mild hypothermia will receive a rapid infusion of 2 liters of 4oC normal saline prior to arrival in the emergency room. Patients randomized to control will receive standard of care following resuscitation from cardiac arrest.
  Other Names: Rapid infusion of cold normal saline
Drug: Rapid infusion of cold normal saline

SUMMARY:
The overall goal of this study is to determine whether initiating hypothermia in cardiac arrest patients as soon as possible in the field results in a greater proportion of patients who survive to hospital discharge compared to standard prehospital/field care.

DETAILED DESCRIPTION:
In this study we will randomize 1,200 cardiac arrest patients who have return of spontaneous circulation (ROSC) to hypothermia with rapid infusion of 2 liters of 4oC Normal Saline IV solution over 20 to 30 minutes, IV sedation and muscle paralysis or to standard of care following ROSC.

The primary objective of this study will be to determine whether induction of mild hypothermia using an infusion of cold normal saline will improve the proportion of patients who survive and are discharged awake from the hospital.

Hypothesis: In cardiac arrest patients who achieve ROSC in the field, initiation of hypothermia by infusion of cold normal saline will result in a greater proportion of cardiac arrest patients discharged awake from the hospital compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* successful resuscitation from out-of-hospital cardiac arrest by paramedics, defined by having a palpable pulse

Exclusion Criteria:

* traumatic cause for cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1359 (Actual)
Dates: Start 2007-12; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Kim, MD, Principal Investigator — University of Washington; Leonard Cobb, MD, Study Director — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Maynard C, Longstreth WT Jr, Nichol G, Hallstrom A, Kudenchuk PJ, Rea T, Copass MK, Carlbom D, Deem S, Olsufka M, Cobb LA, Kim F. Effect of prehospital induction of mild hypothermia on 3-month neurological status and 1-year survival among adults with cardiac arrest: long-term follow-up of a randomized, clinical trial. J Am Heart Assoc. 2015 Mar 11;4(3):e001693. doi: 10.1161/JAHA.114.001693. PMID 25762805
- [Derived] Kim F, Nichol G, Maynard C, Hallstrom A, Kudenchuk PJ, Rea T, Copass MK, Carlbom D, Deem S, Longstreth WT Jr, Olsufka M, Cobb LA. Effect of prehospital induction of mild hypothermia on survival and neurological status among adults with cardiac arrest: a randomized clinical trial. JAMA. 2014 Jan 1;311(1):45-52. doi: 10.1001/jama.2013.282173. PMID 24240712
- [Derived] Ferreira Da Silva IR, Frontera JA. Targeted temperature management in survivors of cardiac arrest. Cardiol Clin. 2013 Nov;31(4):637-55, ix. doi: 10.1016/j.ccl.2013.07.010. PMID 24188226
- [Derived] Soar J, Nolan JP. Mild hypothermia for post cardiac arrest syndrome. BMJ. 2007 Sep 8;335(7618):459-60. doi: 10.1136/bmj.39315.519201.BE. PMID 17823147

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Rapid infusion of 2 liters of 4oC normal saline: Patients randomized to mild hypothermia will receive a rapid infusion of 2 liters of 4oC normal saline prior to arrival in the emergency room. Patients randomized to control will receive standard of care following resuscitation from cardiac arrest.
  Rapid infusion of cold normal saline
- Control: standard of care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 688 | 671
Completed | 688 (5 patients were found to be incarcerated at time of randomization, thus data was not included) | 671
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VF-randomized to Standard Treatment: standard treatment following VF cardiac arrest
- VF-randomized to Hypothermia; Non-VF-randomized to Hypothermia: Rapid infusion of 2 liters of 4oC normal saline: Patients randomized to mild hypothermia will receive a rapid infusion of 2 liters of 4oC normal saline prior to arrival in the emergency room. Patients randomized to control will receive standard of care following resuscitation from cardiac arrest.
  Rapid infusion of cold normal saline
- Non-VF Randomized to Standard Treatment: standard treatment following non-VF cardiac arrest
- Total: Total of all reporting groups
Arm/Group | VF-randomized to Standard Treatment | VF-randomized to Hypothermia | Non-VF Randomized to Standard Treatment | Non-VF-randomized to Hypothermia | Total
Number analyzed (Participants) | 291 | 292 | 380 | 396 | 1359
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (15.6) | 62.1 (14.2) | 67.5 (16.5) | 68.3 (16.3) | 65.1 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 65 | 175 | 180 | 494
  Male | 217 | 227 | 205 | 216 | 865
Region of Enrollment [Number; unit: participants]
  United States | 291 | 292 | 380 | 396 | 1359

OUTCOME MEASURES:

1. Primary Outcome: Number Alive at Hospital Discharge
Time Frame: at hospital discharge
Measure: Number; unit: participants
Arm/Group | VF-randomized to Standard Treatment | VF-randomized to Hypothermia | Non-VF Randomized to Standard Treatment | Non-VF-randomized to Hypothermia
Number analyzed (Participants) | 291 | 292 | 380 | 396
participants | 187 | 183 | 62 | 76

2. Secondary Outcome: Neurologic Status at Discharge-full Recovery
Time Frame: at time of discharge
Measure: Number; unit: participants
Arm/Group | VF-randomized to Standard Treatment | VF-randomized to Hypothermia | Non-VF Randomized to Standard Treatment | Non-VF-randomized to Hypothermia
Number analyzed (Participants) | 291 | 292 | 380 | 396
participants | 145 | 125 | 34 | 36

ADVERSE EVENTS:
Groups:
- Intervention-hypo: Rapid infusion of 2 liters of 4oC normal saline: Patients randomized to mild hypothermia will receive a rapid infusion of 2 liters of 4oC normal saline prior to arrival in the emergency room. Patients randomized to control will receive standard of care following resuscitation from cardiac arrest.
  Rapid infusion of cold normal saline
- Control-standard Care: standard care
Arm/Group | Intervention-hypo | Control-standard Care
Serious Adverse Events (participants affected / at risk) | 547/688 | 513/671
Other Adverse Events (participants affected / at risk) | 0/688 | 0/671
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Intervention-hypo (N=688) | Control-standard Care (N=671)
Re-arrest postrandomization (Cardiac disorders) | 176/686 | 138
Use of pressers post randomization (Cardiac disorders) | 62/686 | 59
prehospital deaths (Cardiac disorders) | 9 | 11
death in emergency dept. (Cardiac disorders) | 88 | 85
use of diuretics first 12 h (Cardiac disorders) | 119/674 | 81/648
pulmonary edema on first chest X-ray (Cardiac disorders) | 256/631 | 184/609

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No